CLINICAL TRIAL: NCT03010657
Title: Dairy Products to Maintain Muscle Mass in People Undergoing Treatment for Lung Cancer
Brief Title: Modifying Your Diet to Support Muscle During Cancer Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA-CC-16-0851; NCT03559881 (obsolete NCT alias)
Record Dates: First submitted 2016-12-20; First posted 2017-01-05 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Skeletal muscle mass; muscle strength; dairy products; high protein diet; cancer treatment; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects will add certain foods to what they normally eat.
  Interventions: Other: Intervention
- Non-experimental intervention (No Intervention): Subjects will continue eating normally.

INTERVENTIONS:
Other: Intervention — Subjects will be asked to consume certain foods during chemotherapy treatment.
  Arms: Intervention

SUMMARY:
In a person with cancer, low muscle mass and strength increases the risks of suffering from severe complications of the disease, its treatment, and dying. To prevent muscle loss in cancer, stimulating muscle protein anabolism (growth) by fueling muscles with protein is crucial. Dairy products are not only a source of high-quality protein but are a preferred food choice for cancer patients as they progress through chemotherapy treatment. Although commercially available oral nutritional supplements containing essential amino acids are often promoted for protein anabolism, these products are not preferred by cancer patients. Moreover, our research group has shown that patients consuming oral nutritional supplements actually lose more weight than those who chose regular whole-food items. Evidence of the health effects of consuming dairy products is needed to influence dietary recommendations for people with cancer. The objective of our study is to perform a clinical trial to evaluate the efficacy of dairy products to maintain muscle mass and strength and improve patient outcomes in people undergoing chemotherapy treatment for cancer.

DETAILED DESCRIPTION:
Muscle wasting is prevalent among cancer patients and cancer treatment can lead to further muscle depletion which is associated with poor outcomes. Dairy products contain complete proteins of high quality and our previous study has shown a preference for dairy products in cancer patients during cancer treatment. This study aims to demonstrate a proof of principle that consumption of a diet high in protein and rich in dairy products will support the maintenance of muscle mass and strength, therefore improving outcomes in cancer patients undergoing treatment.

Methods: The primary outcome is change in muscle mass during cisplatin and/or immunotherapy treatment. Skeletal muscle index was measured by computed tomography (CT). To assess the physical function and muscle strength of patients, short physical performance battery and hand-held dynamometry tests were performed. Patients whose habitual protein intakes were low, received individual dietary instruction from a registered dietician on how to achieve at least one meal per day consisting of a minimum of 30 g of protein derived from at least 50% dairy products as well as 50% of total protein intake from dairy. Patients in a conventional control group continued their habitual dietary intake along with the standard of care. Subjects in the intervention group began consuming their diets immediately after all baseline measurements were collected and continued through treatment, lasting until their follow-up CT scan.

Results: This trial is in progress. It is expected that high protein diet rich in dairy products can maintain patient muscle mass and strength during chemotherapy compared to a low protein diet.

Conclusions: This study will represent a food based nutrition intervention that addresses limiting nutrients to improve outcomes for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of lung cancer scheduled for platinum-based chemotherapy and/or immunotherapy.
* Patients with a computed tomography (CT) image, which includes scans of the 3rd lumbar region, taken within 45 days before initiation of chemotherapy and/or immunotherapy.
* Ability to maintain oral intake.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2 / Karnofsky Performance Status between 60-100.
* Ability to give written, informed consent.

Exclusion Criteria:

* Co-morbidities that would be expected to interfere with the primary outcome measure (e.g. neuromuscular diseases).
* Patients on long term drugs or supplements that modify muscle metabolism (e.g. corticosteroids, anti-androgens, omega-3 fatty acids).
* Life expectancy <3 months.
* Severe food restriction(s) (e.g. food allergy, intolerance or dietary pattern) that would inhibit the study intervention food modification.
* An inability to comply with study instructions.
* Patients engaged in a total of ≥50 minutes of moderate-to-vigorous cardiovascular exercise per week and/or structured resistance exercise occurring ≥2 times per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in muscle mass | 12 weeks
  CT-derived changes in muscle mass occurring during the course of chemotherapy and/or immunotherapy treatment

SECONDARY OUTCOMES:
Change in muscle strength | Baseline
  Hand grip
Change in muscle strength | 10 weeks
  Hand grip
Change in physical performance | Baseline
  Short physical performance battery protocol
Change in physical performance | 10 weeks
  Short physical performance battery protocol
Change in quality of life | Baseline
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (30 and LC13)
Change in quality of life | 10 weeks
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (30 and LC13)
Change in nutritional status | Baseline
  Patient Generated Subjective Global Assessment
Change in nutritional status | 10 weeks
  Patient Generated Subjective Global Assessment
Change in inflammatory status | Baseline
  C-reactive protein/albumin ratio
Change in inflammatory status | 10 weeks
  C-reactive protein/albumin ratio

CONTACTS AND LOCATIONS:
Overall Officials: Vera Mazurak, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada